CLINICAL TRIAL: NCT06964321
Title: Effectiveness of Intercostal Tube Drainage Vs Pigtail Catheter Drainage Vs Ultrasound-Guided Aspiration in Management of Massive Malignant Pleural Effusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mark Badrat William Mansour, residant doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IT drainage-pigtail-US Aspirat
Record Dates: First submitted 2025-05-01; First posted 2025-05-09 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Active Comparator): intercostal tube drainage in managing massive malignant pleural effusion (MPE).
  Interventions: Procedure: intercostal tube drainage
- Group B (Active Comparator): big tail catheter drainage in managing massive malignant pleural effusion (MPE).
  Interventions: Procedure: big tail catheter drainage
- Group C (Active Comparator): ultrasound-guided aspiration in managing massive malignant pleural effusion (MPE).
  Interventions: Procedure: ultrasound-guided aspiration

INTERVENTIONS:
Procedure: intercostal tube drainage — intercostal tube drainage in managing massive malignant pleural effusion (MPE).
  Arms: Group A
Procedure: big tail catheter drainage — big tail catheter drainage in managing massive malignant pleural effusion (MPE).
  Arms: Group B
Procedure: ultrasound-guided aspiration — ultrasound-guided aspiration in managing massive malignant pleural effusion (MPE).
  Arms: Group C

SUMMARY:
Pleural effusion is common in different diseases and especially malignant effusions can have fast onset symptoms such as chest pain, dyspnoea, and coughing. Malignant pleural effusion (MPE) is an exudative effusion with malignant cells.

It is a common symptom and accompanying presentation of metastatic disease. It Impacts up to 15% of all patients with cancer and is the most common in breast, lung, cancer, lymphoma, and gynaecological malignancies . There are 150,000 new cases of MPE in the United States yearly and 100,000 in Europe . Patients have an overall survival (OS) rate of 3-12 months after the initial diagnosis . Malignant pleural effusion (MPE) poses significant challenges in management, impacting patient quality of life and overall prognosis. Almost all radiological procedures can help diagnose pleural effusions . Thoracentesis is used as a diagnostic and therapeutic tool. The procedure has been modified with the addition of ultrasound, that is very functional for targeting certain anatomical areas of the pleura and finding an appropriate entry point . Three primary strategies are commonly employed: intercostal tube drainage, big tail catheter drainage, and ultrasound-guided aspiration. This study aims to evaluate these methods' efficacy, safety, and outcomes. To compare intercostal tube drainage, big tail catheter drainage, and ultrasound-guided aspiration in managing massive malignant pleural effusion (MPE).

ELIGIBILITY:
Inclusion Criteria:

* Adult patient aged 18 years old and above.
* Patients diagnosed with massive malignant pleural effusion (MPE) requiring intervention.

Exclusion Criteria:

* Pediatric patients aged below 18 years
* Patients with non-malignant causes of pleural effusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Resolution of Pleural Effusion | baseline
  Resolution of Pleural Effusion: Defined as complete or partial resolution based on imaging studies (e.g., chest X-ray or ultrasound).